CLINICAL TRIAL: NCT02561767
Title: The Efficacy and Safety of Bone Marrow-derived Mesenchymal Stem Cells in Kidney Transplantation From Chinese Donation After Citizen Death (DCD): A Multi-center Randomized Controlled Trial
Brief Title: Effect of BM-MSCs in DCD Kidney Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Changxi Wang, Director of Organ Transplant Center, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSCs-KTx-DCD-150924
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Transplantation; Acute Kidney Tubular Necrosis
Keywords: kidney transplantation; mesenchymal stem cell; donation after citizen's death; ischemia reperfusion injury; renal function recovery
MeSH Terms: conditions — Kidney Tubular Necrosis, Acute; Reperfusion Injury | interventions — Sodium Chloride; Neoadjuvant Therapy; Basiliximab; Maintenance; cni protein, Drosophila; Steroids; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSCs group (Experimental): Allogeneic bone marrow-derived mesenchymal stem cells (10^6/kg) from third party donors is intravenously given at day 0 (after renal artery reperfusion), day 7, day 14 and day 21.Induction therapy: ATG or Basiliximab; Maintenance therapy: low-dose Tacrolimus + mycophenolic acid + prednisone.
  The third-party MSCs have no similar HLA alleles of kidney donors, and have no HLA alleles specific to preformed anti-HLA antibodies in recipients prior to KTx.
  Interventions: Other: bone marrow-derived mesenchymal stem cells; Drug: Induction therapy (ATG or Basiliximab); Drug: Maintenance therapy (Low-dose CNI + MPA + steroids)
- Control group (Placebo Comparator): Placebo (saline) is intravenously given at day 0 (after renal artery reperfusion), day 7, day 14 and day 21. Induction therapy: ATG or Basiliximab; Maintenance therapy: low-dose Tacrolimus + mycophenolic acid + prednisone.
  Interventions: Other: Saline; Drug: Induction therapy (ATG or Basiliximab); Drug: Maintenance therapy (Low-dose CNI + MPA + steroids)

INTERVENTIONS:
Other: bone marrow-derived mesenchymal stem cells — BM-MSCs is harvested from third-party health volunteer donors.
  Other Names: BM-MSCs
  Arms: MSCs group
Other: Saline — Saline as placebo of MSCs
  Arms: Control group
Drug: Induction therapy (ATG or Basiliximab) — ATG, antithymocyte globulin; Basiliximab, anti-CD25 mAb. Recipients receive ATG or Basiliximab as induction therapy in both MSCs group and control group.
  Other Names: ATG or Basiliximab
Drug: Maintenance therapy (Low-dose CNI + MPA + steroids) — Maintenance immunosuppressive therapy consists of low-dose tacrolimus and mycophenolic acid and steroids. Recipients receive the same maintenance therapy in both MSCs group and control group.
  Other Names: Low-dose tacrolimus + Mycophenolic acid (MPA) + steroids

SUMMARY:
This study is designed to determine the efficacy and safety of allogeneic bone marrow-derived mesenchymal stem cells in kidney transplantation from Chinese donation after citizen's death (DCD). A pair uremia patients receiving kidney grafts from a same donor are randomized into two groups: MSCs group and control group. Besides routine induction therapy (ATG or Basiliximab) and maintenance immunosuppressive drugs (low-dose Tacrolimus + MPA + prednisone), patients in MSCs group are administered MSCs treatment (1*10^6/kg). Allogeneic bone marrow-derived MSCs (1*10^6/kg) are given intravenously at day 0 (post renal reperfusion during surgery), day 7, day 14 and day 21. The renal allograft function, rejection, patient/graft survival and severe adverse events within 12 months post-transplant are monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Primary kidney transplantation
2. Receiving induction therapy and combined immunosuppressive regimens (CNIs + MPA + steroids)
3. Patient is willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months

Exclusion Criteria:

1. Secondary kidney transplantation
2. Combined or multi-organ transplantation
3. Women who are pregnant, intend to become pregnant in the next 1 years, breastfeeding, or have a positive pregnancy test on enrollment or prior to study medication administration
4. Panel reactive antibody (PRA)>20%
5. CDC crossmatch is positive
6. Donors or recipients are known hepatitis C antibody-positive or polymerase chain reaction (PCR) positive for hepatitis C
7. Donors or recipients are known hepatitis B surface antigen-positive or PCR positive for hepatitis B
8. Donors or recipients are known human immunodeficiency virus (HIV) infection
9. Patients with active infection
10. Recipients with a history of substance abuse (drugs or alcohol) within the past 6 months, or psychotic disorders that are not capable with adequate study follow-up.
11. Patients with severe cardiovascular dysfunction
12. WBC<3*10^9/L or RBC <5g/dL
13. Highly allergic constitution or having severe history of allergies.
14. Patients with active peptic ulcer disease, chronic diarrhea, or gastrointestinal problem affect absorption
15. Patients with a history of cancer within the last 5 years
16. Prisoner or patients compulsorily detained (involuntarily incarcerated) for treatment or either a psychiatric or physical (e.g. infectious disease) illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate | 1 month
  eGFR at one month post-transplant

SECONDARY OUTCOMES:
Incidence of slow graft function | 12 months
Incidence of delayed graft function | 12 months
Proportion of normal renal function recovery | 12 months
Time to renal function recovery | 12 months
Patient survival | 12 months
Renal graft survival | 12 months
Incidence of acute rejection | 12 months
Severe adverse events | 12 months
Estimated glomerular filtration rate | 12 months
  eGFR up to 12 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Changxi Wang, M.D., Ph.D, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Peng Y, Ke M, Xu L, Liu L, Chen X, Xia W, Li X, Chen Z, Ma J, Liao D, Li G, Fang J, Pan G, Xiang AP. Donor-derived mesenchymal stem cells combined with low-dose tacrolimus prevent acute rejection after renal transplantation: a clinical pilot study. Transplantation. 2013 Jan 15;95(1):161-8. doi: 10.1097/TP.0b013e3182754c53. PMID 23263506
- See also: Previous publication — http://www.ncbi.nlm.nih.gov/pubmed/23263506